CLINICAL TRIAL: NCT03871959
Title: CATRIPCA - A Phase I Study of PD1 Monoclonal Antibody (Pembrolizumab) In Combination With a IAP Antagonist (Debio 1143) In (Exocrine) Pancreatic And Colorectal Non MSI-high Advanced/Metastatic Adenocarcinoma.
Brief Title: Pembrolizumab In Combination With Debio 1143 In Pancreatic and Colorectal Advanced/Metastatic Adenocarcinoma
Acronym: CATRIPCA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Debiopharm International SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ET16-023 CATRIPCA
Record Dates: First submitted 2019-03-08; First posted 2019-03-12 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Adenocarcinoma of the Pancreas; Adenocarcinoma of the Colon; Adenocarcinoma of the Rectum
Keywords: PD1 Monoclonal Antibody; IAP Antagonist; phase I; MSI
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — pembrolizumab; N-benzhydryl-5-(2-(methylamino)propanamido)-3-(3-methylbutanoyl)-6-oxodecahydropyrrolo(1,2-a)(1,5)diazocine-8-carboxamide

STUDY DESIGN:
Intervention Model Description: The dose escalation part will follow a classical 3+3 design. 3 to 6 patients will be enrolled at each Dose Level depending of the number of Dose Limiting Toxicities observed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab + Debio 1143 (Experimental): Pembrolizumab : 200 mg, intravenous (IV), to be administered on Day 1 of every 3-week cycle i.e. Q3W.
  Debio 1143 : 3 escalating dose level (100 mg, 150 mg, 200 mg) administered daily for 14 days over a 21-day cycle period.
  Interventions: Drug: Pembrolizumab; Drug: DEBIO1143

INTERVENTIONS:
Drug: Pembrolizumab — 200 mg, intravenous (IV), to be administered on Day 1 of every 3-week cycle i.e. Q3W.
  Other Names: Keytruda
Drug: DEBIO1143 — 3 escalating dose level (100 mg, 150 mg, 200 mg) of Debio 1143 administered daily for 14 days over a 21-day cycle period.

SUMMARY:
This trial is a Phase I study to be conducted in patients with non-MSI-high advanced/metastatic pancreatic ductal adenocarcinoma (PDAC) or colorectal cancer (CRC) and is divided in two Parts.

* Dose escalation Part :To determine the Maximum Tolerated Dose (MTD) and the Recommended Dose for Phase 2 (RP2D) of Debio1143 when combined with a fixed dose of Pembrolizumab.
* Extension Part: To evaluate preliminary efficacy data of the proposed combination.

DETAILED DESCRIPTION:
All patient wil receive a combinaison of Pembrolizumab and Debio 1143. Pembrolizumab is a potent and highly selective humanized monoclonal antibody (mAb) of the IgG4/kappa isotype designed to directly block the interaction between PD-1 and its ligands, PD-L1 and PD-L2.

Debio 1143 is an investigational, oral monovalent second mitochondrial-derived activator of caspases (SMAC) mimetic designed to promote programmed cell death (apoptosis) in tumor cells and anti-tumour immunity. By antagonizing the activity of inhibitor of apoptosis proteins (IAPs (X-linked IAP [XIAP], cellular IAP 1 [cIAP1], cellular IAP 2 [cIAP2] and melanoma-linked IAP [ML-IAP])), Smac mimetics are an interesting treatment approach for cancer that may foster better tumor responses to chemo/radiotherapy- and/or immuno-therapy.

A Dose escalation part (n= up to 18 patients ) aiming to define the Maximum Tolerated Dose and the the Recommended Dose for Phase 2 of the proposed combination. A classical 3+3 design will be used with a fixed dose of Pembrolizumab (200 mg, intravenous , to be administered on Day 1 of every 3-week cycle i.e. Q3W) and 3 escalating dose level of Debio 1143 administered daily for 14 days over a 21-day cycle period.

There will be a 24-hour delay between the first and subsequent patients enrolled in each DL cohort to maximize the safety of enrolled patients.

An extension part (n=28 patients: 14 patients per cohort) aiming to evaluate the clinical activity of the proposed combination.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged of at least 18 years on day of signing informed consent.
* Histologically-confirmed diagnosis of Stage III or IV (according to the current version of the American Joint Committee on Cancer (AJCC)) of PDAC or Stage IV CRC.

Note: pancreatic endocrine tumors are not eligible.

* Previous treatment in the metastatic / advanced stage: PDAC: at least one line of chemotherapy and CRC: at least one line of chemotherapy containing 5-FU, oxaliplatin, irinotecan, plus bevacizumab if patient is eligible, plus anti-EGFR if CRC with RAS wild-type.
* Documented radiological disease progression as per RECIST V1.1 at time of inclusion.
* At least one measurable lesion according to RECIST v1.1.
* Presence of at least one tumor lesion with a diameter ≥20 mm, visible by medical imaging and accessible to repeatable percutaneous (needle biopsies 18 gauge or larger) sampling that permit core needle biopsy (ideally 4 cores) without unacceptable risk of a major procedural complication.

Note: 1. endoscopic biopsies are not allowed. 2. Lymph nodes, lung and RECIST target lesions are not suitable for de novo biopsies.

- Availability of a representative formalin-fixed and paraffin-embedded (FFPE) primary and/or metastatic tumor tissue with an associated pathology report.

Note: Fine needle aspirates, and bone biopsies do not satisfy the requirement for tumor tissue.

Note : If adequate tissue from distinct timepoints (such as time of initial diagnosis and time of disease recurrence and/or multiple metastatic tumors is available), priority should be given to the tissue most recently collected (ideally subsequent to the most recent systemic therapy).

* ECOG Performance Status (PS) 0 or 1 (See Appendix 1).
* Life expectancy of at least 12 weeks.
* Demonstrate adequate organ function as defined in table below, all screening laboratory tests should be performed within 7 days prior C1D1.

HEMATOLOGICAL Absolute neutrophil count (ANC) ≥ 1.5 G/L Platelets ≥ 100 G/L Hemoglobin ≥ 9 g/dL (without transfusion within 7 days) RENAL Serum creatinine OR Creatinine clearance according to CKD-EPI ≤ 1.5 × Upper Limit of Normal (ULN) OR ≥ 50 mL/min/1.73m2 HEPATIC Serum total bilirubin ≤ 1.5 × ULN (except for patients with Gilbert disease for whom a total serum bilirubin ≤ 3 x ULN is acceptable). OR Direct bilirubin ≤ ULN for patients with total bilirubin levels > 1.5 × ULN ASAT and ALAT ≤ 3 × ULN (or ≤ 5 × ULN in case of liver metastasis or hepatic infiltration) COAGULATION INR and Activated Partial Thromboplastin Time (aPTT) ≤ 1.5 × ULN Note: This is applicable only for patients not receiving an anticoagulant treatment: patients receiving therapeutic anticoagulation must be on stable dose.

* Able to swallow and retain orally administered medication.
* Minimal wash-out period for the following treatments (= minimal delay between the last dose of these treatments and C1D1): Chemotherapy, tyrosine kinase inhibitor or radiation therapy : 2 weeks; Immunosuppressive medication: 4 weeks, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid; Any investigational agents: 5 half-lives of the investigation agent with a minimum of 2 weeks; Monoclonal antibodies: 4 weeks; Major surgical procedure, open biopsy (excluding skin cancer resection or screening biopsy), or significant traumatic injury : 2 weeks; Live vaccines : 4 weeks.
* Women of child-bearing potential must have a negative serum pregnancy test at Screening and must agree to use 2 effective forms of contraception from the time of the negative pregnancy test up to 120 days after the last dose of study drugs.
* Fertile men must agree to use contraceptive measures up to 120 days after the last dose of study drugs.
* Patients who understand, sign, and date the written voluntary informed consent form at the screening visit prior to any protocol-specific procedures. Patient should be able and willing to comply with study visits and procedures as per protocol.
* Patients must be covered by a medical insurance.

Exclusion Criteria:

* Patients amenable to therapy with curative intent.
* Patient participating to another clinical trial with a medicinal product.
* Patients with microsatellite instability (MSI)-high or mismatch repair MMR-deficient tumors.
* Patients who have not recovered from adverse events (i.e. > Grade 1 according to NCI CTCAE v5.0 See Appendix 5) due to prior treatment with anti-cancer agents with exception of Grade 2 neuropathy, any Grade alopecia or lab values presented in criteria I10.
* Patients who have received prior therapy with an anti-PD-1, anti-PD-L1, anti-CTL-A4 and any ICIs or IAP inhibitors.
* Patients who have a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
* Patients with known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to C1D1 and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids (at doses higher than 10 mg/d of methylprednisolone or equivalent) for at least 4 weeks prior C1D1.
* Patients with a history of autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids (at doses higher than 10 mg/d of methylprednisolone or equivalent) or immunosuppressive agents.
* Patients with history of (non-infectious) pneumonitis that required steroids, evidence of interstitial lung disease or active, non-infectious pneumonitis.
* Patients with an evidence of active infection requiring systemic therapy.
* Patients with a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial.
* Patients with a history of uncontrolled or symptomatic, clinically significant cardiovascular disease : stroke, myocardial infarction, angina pectoris, arrhythmias, congestive heart failure (NYHA Class >2), or myocarditis within 6 months prior to first study drug administration.
* Patient with a history of organ transplant including stem cell allograft.
* Patients receiving or to be treated during the treatment period with one of the following forbidden treatment: Any anti-cancer systemic chemotherapy, targeted therapy or biological therapy including any immunotherapy not mentioned in this protocol; Any investigational agents other than Debio-1143; Radiation therapy; Live vaccines, Major surgery; Corticosteroids for any purpose other than to modulate symptoms from an event of clinical interest of suspected immunologic etiology. The use of physiologic doses of corticosteroids may be approved after consultation with the sponsor; Strong P-gp inhibitors or inducers.
* Patients with hypersensitivity to Pembrolizumab or any of its excipients.
* Patients with a known history of active TB (Bacillus Tuberculosis).
* Patients with : Active hepatitis B (chronic or acute; defined as having a positive hepatitis B surface antigen [HBsAg] test at screening), or Active hepatitis C. Patients positive for hepatitis C virus (HCV) antibody are eligible only if PCR is negative for HCV RNA, or HIV infection.
* Patients with known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Patients who are pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-06-08 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 21 days
  To determine the Maximum Tolerated Dose of Debio1143 when combined with a fixed dose of Pembrolizumab.
Recommended Dose for Phase 2 | 21 days
  To determine the Recommended Dose for Phase 2 (RP2D) of Debio1143 when combined with a fixed dose of Pembrolizumab.
Extension Part Objective Response Rate | 12 weeks
  The Objective Response Rate will be defined as the proportion of patients with complete response or partial response, as per RECIST V1.1.

SECONDARY OUTCOMES:
Duration of response | Up to 2 years
  The duration of response will be measured from the time of first documented response (Complete Response or Partial Response as per RECIST V1.1) until the first documented disease progression or death due to underlying cancer, and censored at the date of the last available tumor assessment.
Clinical Benefit Rate | 12 weeks
  The Clinical Benefit Rate will be defined as the proportion of patients with Complete Response, Partial Response or stable disease according to RECIST V1.1.
Tumor-response efficacy 1 | Up to 2 years
  The tumor-response efficacy endpoints described above will be evaluated by investigator-assessed RECIST v1.1 (Eisenhauer et al. E J Cancer 2009).
Tumor-response efficacy 2 | Up to 2 years
  The tumor-response efficacy endpoints described above will be evaluated by modified criteria for immunotherapies iRECIST (Seymour et al. Lancet Oncol 2017).
Progression-Free Survival | Up to 2 years
  Progression-Free Survival (PFS) will be measured from the C1D1 until the date of event defined as the first documented progression or death from any cause. Patients with no event at the time of the analysis will be censored at the date of the last available tumor assessment.
Overall survival | Up to 2 years
  Overall survival (OS) will measured from C1D1 to the date of death from any cause. Patients who are alive at the time of analysis will be censored at the date of the last contact.
Assessment of safety will be based mainly on the frequency of adverse events based on the common toxicity criteria (CTCAE v5.0) grade | Up to 2 years
  The assessment of safety will be based mainly on the frequency of adverse events based on the common toxicity criteria (CTCAE v5.0) grade.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe CASSIER, MD, Principal Investigator — Centre Leon Berard
Locations (1):
- Centre Léon Bérard, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Crawford N, Stott KJ, Sessler T, McCann C, McDaid W, Lees A, Latimer C, Fox JP, Munck JM, Smyth T, Shah A, Martins V, Lawler M, Dunne PD, Kerr EM, McDade SS, Coyle VM, Longley DB. Clinical Positioning of the IAP Antagonist Tolinapant (ASTX660) in Colorectal Cancer. Mol Cancer Ther. 2021 Sep;20(9):1627-1639. doi: 10.1158/1535-7163.MCT-20-1050. Epub 2021 Aug 13. PMID 34389694